CLINICAL TRIAL: NCT01610427
Title: Optimizing the Quality of Samples Used for the Evaluation of Cell-mediated Immune (CMI) Responses in Antiretroviral Therapy (ART)-naïve Human Deficiency Virus Type 1 (HIV-1)-Infected Subjects
Brief Title: Study to Optimize the Quality of Samples for Cell-mediated Immunity (CMI) in ART-naïve HIV-1-infected Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 116329
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: AIDS; AIDS Vaccines
Keywords: CMI; Antiretroviral therapy-naïve; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

ARMS (1):
- HIV-1 Group (Experimental): Antiretroviral Therapy-naïve HIV1-infected subjects, aged 18 to 55 years, from whom samples for cell-mediated immunity (CMI) were collected. No investigational vaccine was administered.
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — Blood samples will be collected in all subjects at two time points, at the Screening Visit (Day 0) and at the Sample Collection Visit (Day 15)

SUMMARY:
The purpose of this study is to investigate a combined set of parameters deemed to impact the quality of CMI analyses in terms of the proportion of viable lymphocytes in antiretroviral therapy-naïve HIV-1 infected subjects.

DETAILED DESCRIPTION:
This study will address the respective and combined impact of (i) timing between blood collection and peripheral blood mononuclear cells (PBMC) processing ["time-to-process"] and (ii) timing of PBMC resting before stimulation ["resting -time"].

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy all the following criteria at study entry:

* Subjects who the Investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to any study procedure.
* A male or female between and including 18 and 55 years of age at the time of enrollment.
* Confirmed HIV-1 infection.
* ART-naïve and not eligible for ART treatment as per established guidelines. Subjects must never have received ART after HIV diagnosis, including lamivudine used for chronic hepatitis B infection. The exception to this is short-term ART for prevention of mother-to-child transmission (PMTCT) which must have been completed at least 360 days prior to enrollment.
* Viral load level between and including 2,000 and 100,000 copies/mL at screening.
* CD4+ T cell count >500 cells/mm3 at screening.
* If the subject is female, she must be of non-childbearing potential, i.e., have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal. Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at screening, and
  * has agreed to continue adequate contraception during the entire study period.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any exclusion criterion applies, the subject must not be included in the study:

* Infection with HIV-2. This includes subjects with dual infection with HIV-1/HIV-2.
* Planned use of any hematotoxic product during the study period.
* Planned use of any investigational or non-registered product during the study period.
* Acute or chronic, clinically relevant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination, serology and/or medical history at screening.
* Grade 3 or grade 4 laboratory abnormalities, as defined by Division of AIDS (DAIDS) grading table, at screening.
* Any condition which, in the opinion of the Investigator, could compromise the subject's adherence to the study protocol.
* Planned administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the Sample Collection Visit (Visit 2). Vaccine can be administered as after sampling in Visit 2.
* Pregnant or lactating female.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2012-10-30 (Actual); Study Completion 2012-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourguignon P, Clement F, Renaud F, Le Bras V, Koutsoukos M, Burny W, Moris P, Lorin C, Collard A, Leroux-Roels G, Roman F, Janssens M, Vandekerckhove L. Processing of blood samples influences PBMC viability and outcome of cell-mediated immune responses in antiretroviral therapy-naive HIV-1-infected patients. J Immunol Methods. 2014 Dec 1;414:1-10. doi: 10.1016/j.jim.2014.09.001. Epub 2014 Sep 16. PMID 25224748

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 31 subjects registered in the study, 9 subjects were screen failures and 22 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | HIV-1 Group
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African heritage / African American | 1
  Race: Asian - East Asian heritage | 1
  Race: White - Caucasian / European heritage | 20

OUTCOME MEASURES:

1. Primary Outcome: Lymphocytes Viability Prediction (LOGIT Transformed) in CMI Samples Post-overnight Incubation Time Before Intracellular Cytokine Staining (ICS): "Intercept" Parameter Estimate of the Prediction Model - Condition "None" Resting Time Not Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=2h, 6h or 18h ["none" resting time not included]) conditions to select the best combination of these two parameters to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10^P/(1 + 10^P)*100 with P for Prediction.The optimum of the viability was predicted as P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + a*a*TP*TP + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the 3 first primary outcomes. And a and b are log-transformed parameters corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting the intercept i.e. expected mean value of Prediction when "TP" and "RT" = 0. The optimum of this Design of Experiment is presented in outcome 4.
Time Frame: At Day 15 (sample collection visit)
Population: The analysis was performed on the According to Protocol (ATP) Sample Collection cohort, which included all subjects accepted into the analysis.
Measure: Log Mean (Standard Error); unit: Unitless assessment of prediction
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Unitless assessment of prediction | 0.6490 (0.06989)

2. Primary Outcome: Lymphocytes Viability Prediction (LOGIT Transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: Time to Process and Resting Time Parameter Estimates of the Prediction Model - Condition "None" Resting Time Not Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=2h, 6h or 18h ["none" resting time not included]) conditions to select the best combination of these two parameters to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction.The optimum of the viability was predicted as P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + a*a*TP*TP + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the 3 first primary outcomes. And a and b are log-transformed parameters corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting "TP" and "RT" estimates expressed as log(hours). The optimum of this Design of Experiment (DOE) is presented in outcome 4.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Log(hours)
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Log(hours)
  TP | 0.1724 (0.1152)
  RT | 0.9578 (0.1342)

3. Primary Outcome: Lymphocytes Viability Prediction (LOGIT Transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: TP*RT, TP*TP and RT*RT Parameter Estimates of the Prediction Model - Condition "None" Resting Time Not Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=2h, 6h or 18h ["none" resting time not included]) conditions to select the best combination of these two parameters to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction.The optimum of the viability was predicted as P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + a*a*TP*TP + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the 3 first primary outcomes. And a and b are log-transformed parameters corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting TP*RT, TP*TP and RT*RT estimates expressed as log(hours^2). The optimum of this DOE is presented in outcome 4.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Log(hours^2)
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Log(hours^2)
  TP*RT | 0.1120 (0.05041)
  TP*TP | -0.2934 (0.06426)
  RT*RT | -0.9364 (0.08133)

4. Primary Outcome: Lymphocytes Viability Prediction (LOGIT Transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: Optimum Mean Cell Viability Estimate by the Prediction Model - Condition "None" Resting Time Not Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=2h, 6h or 18h ["none" resting time not included]) conditions to select the best combination of these two parameters to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction.The optimum of the viability was predicted as P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + a*a*TP*TP + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the 3 first primary outcomes. And a and b are log-transformed parameters corresponding respectively to the "TP" and the "RT" where the prediction has to be done. The optimum predicted mean cell viability of this Design of Experiment is presented in this outcome and expressed as percentage.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Number; unit: Percentage of viable lymphocytes
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Percentage of viable lymphocytes | 89.69

5. Primary Outcome: Lymphocytes Viability Prediction (Non-transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: "Intercept" Parameter Estimate of the Prediction Model - Condition "None" Resting Time Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=0h) conditions in order to select the best combination of these two parameters with the aim to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction. The optimum of the viability was predicted as follows. P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the primary outcomes 5, 6 and 7. And "a" and "b" are parameters (hour) corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting the intercept i.e. expected mean value of Prediction when "TP" and "RT" = 0. The optimum of this Design of Experiment is presented in outcome 8.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Unitless assessment of prediction
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Unitless assessment of prediction | 0.8145 (0.03753)

6. Primary Outcome: Lymphocytes Viability Prediction (Non-transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: Time to Process and Resting Time Parameter Estimates of the Prediction Model - Condition "None" Resting Time Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=0h) conditions in order to select the best combination of these two parameters with the aim to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction. The optimum of the viability was predicted as follows. P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the primary outcomes 5, 6 and 7. And "a" and "b" are parameters (hour) corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting "TP" and "RT" estimates expressed as log(hours). The optimum of this Design of Experiment (DOE) is presented in outcome 8.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Log(hours)
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Log(hours)
  TP | -0.01853 (0.001194)
  RT | 0.04616 (0.005642)

7. Primary Outcome: Lymphocytes Viability Prediction (Non-transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: TP*RT and RT*RT Parameter Estimates of the Prediction Model - Condition "None" Resting Time Included
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=0h) conditions in order to select the best combination of these two parameters with the aim to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction. The optimum of the viability was predicted as follows. P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the primary outcomes 5, 6 and 7. And "a" and "b" are parameters (hour) corresponding respectively to the "TP" and the "RT" where the prediction has to be done. This outcome is presenting TP*RT and RT*RT estimates expressed as log(hours^2). The optimum of this DOE is presented in outcome 8.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Log Mean (Standard Error); unit: Log(hours^2)
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Log(hours^2)
  TP*RT | 0.000588 (0.000121)
  RT*RT | -0.00367 (0.000284)

8. Primary Outcome: Lymphocytes Viability Prediction (Non-transformed Estimate) in CMI Samples Post-overnight Incubation Time Before ICS: Optimum Mean Cell Viability Estimates by the Prediction Model -Condition "None" Resting Time Included.
Description: The objective was to model lymphocyte viability according to "time-to-process" (TP=2h, 7h or 24h) and "resting time" (RT=0h) conditions in order to select the best combination of these two parameters with the aim to maximize the post-ICS viability in CMI samples collected from ART-naïve HIV-1-infected subjects. Viability (%) = 10 ^ P / (1 + 10 ^ P) * 100 with P for Prediction. The optimum of the viability was predicted as follows. P (LOGIT)= intercept + a*TP + b*RT + a*b*TP*RT + + b*b*RT*RT. Where "intercept", "TP", "RT", "TP*RT", "TP *TP", "RT*RT" are the parameters evaluated and presented in the primary outcomes 5, 6 and 7. And "a" and "b" are parameters (hour) corresponding respectively to the "TP" and the "RT" where the prediction has to be done. The optimum predicted mean cell viability of this Design of Experiment is presented in this outcome and expressed as percentage.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Number; unit: Percentage of viable lymphocytes
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Percentage of viable lymphocytes | 89.49

9. Secondary Outcome: Percentage of Viable Lymphocytes in the CMI Samples, Post-overnight Incubation (Classic) Before ICS and Post-6 Hour Incubation Before ICS
Description: The percentage of viable lymphocytes was determined by Forward Scatter/Side Scatter (FSC/SSC) and LIVE/DEAD gating during flow cytometry analysis for each incubation of time-to-time process (TP) = 2h, 7h and 24 h and resting time (RT) = 18h for the comparison of resting time = 18h and classic incubation time versus resting time = 18h and post-6h incubation time.
Time Frame: A Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of viable lymphocytes
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Percentage of viable lymphocytes
  TP=2h; RT=18h; post 6h incubation | 82.30 [79.57 to 84.74]
  TP=2h; RT=18h; classic incubation | 72.72 [69.07 to 76.09]
  TP=7h; RT=18h; post 6h incubation | 82.49 [76.09 to 84.97]
  TP=7h; RT=18h; classic incubation | 73.65 [70.00 to 77.01]
  TP=24h; RT=18h; post 6h incubation | 72.64 [68.83 to 76.15]
  TP=24h; RT=18h; classic incubation | 64.60 [60.41 to 68.58]

10. Secondary Outcome: Magnitude of HIV-1 RT Specific Cluster of Differentiation 40 Ligand (CD40L+) CD4+ T Cell Responses in the CMI Samples Post-overnight ICS/Post 6 Hour ICS, Expressing at Least One Cytokine
Description: Data were collected but could not be reported as data were below level of detection.
Time Frame: At Day 15 (sample collection visit)
Population: The analysis was to be performed on the According to Protocol (ATP) Sample Collection cohort. Data were collected but could not be reported as data were below the detection level.
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 0

11. Secondary Outcome: Magnitude of HIV-RT Specific (Background Reduced) CD8+ T Cell Responses in the CMI Samples Post-overnight ICS/Post 6 Hour ICS, Expressing at Least One Cytokine
Description: HIV-RT specific responses of CD8+ T cells expressing at least one cytokine, among: Interleukin-2 (IL-2), Interferon-gamma (IFN-g) and Tumor necrosis factor alpha (TNF-a),after stimulation with HIV-1 peptide pools for time-to-process (TP) (2, 7, 24 hours) and resting time (RT) (0,2,6,18 hours) post-overnight ICS and for time-to-process (7 hours) and resting time (18 hours) post 6 hours ICS.
Time Frame: At Day 15 (sample collection visit)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of CD8+ T cells
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Percentage of CD8+ T cells
  TP 2h RT 0h post-overnight ICS | 0.257075 [0.165275 to 0.492275]
  TP 2h RT 2h post-overnight ICS | 0.2757 [0.193275 to 0.56075]
  TP 2h RT 6h post-overnight ICS | 0.3059 [0.122015 to 0.465168]
  TP 2h RT 18h post-overnight ICS | 0.3114 [0.1855 to 0.946325]
  TP 7h RT 0h post-overnight ICS | 0.23485 [0.10595 to 0.44535]
  TP 7h RT 2h post-overnight ICS | 0.2761 [0.16446 to 0.54085]
  TP 7h RT 6h post-overnight ICS | 0.2615 [0.141975 to 0.6853]
  TP 7h RT 18h post-overnight ICS | 0.35455 [0.220358 to 0.8207]
  TP 7h RT 18h post 6h ICS | 0.117 [0.0729 to 0.29695]
  TP 24h RT 0h post-overnight ICS | 0.18731 [0.130225 to 0.43595]
  TP 24h RT 2h post-overnight ICS | 0.29285 [0.141575 to 0.644325]
  TP 24h RT 6h post-overnight ICS | 0.2496 [0.1472 to 0.7351]
  TP 24h RT 18h post-overnight ICS | 0.3663 [0.2138 to 1.0977]

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitali-zation or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the whole study period (From Day 0 to Day 15)
Population: The analysis was performed on the Total eligible cohort which included all subjects in the Total cohort (all enrolled subjects) who fulfilled eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-1 Group
Number analyzed (Participants) | 22
Participants | 0

ADVERSE EVENTS:
Time Frame: SAEs: during the whole study period (From Day 0 to Day 15)
Description: Only All-Cause Mortality and Serious Adverse Events were assessed. Other (Not Including Serious) Adverse Events were not monitored during this study period.
Arm/Group | HIV-1 Group
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.